CLINICAL TRIAL: NCT00935896
Title: Mechanical Ventilation With High Tidal Volume Induces Inflammation In Patients Without Lung Disease
Brief Title: High Tidal Volume Induces Inflammation In Normal Lungs
Acronym: Normallung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Programa de Pós-Graduação em Clínica Médica (Unknown); Faculdade de Medicina (Ambiguous)
Responsible Party: Prof. Gilberto Friedman, Faculdade de Medicina - Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: normal lung - V1; CAPES-PROF - UFRGS
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Mechanically Ventilated Patients; Normal Lungs
Keywords: Ventilator-associated lung injury; Tumor necrosis factor-alpha; Interleukin-8; Mechanical ventilation; Low tidal volume ventilation; Normal lungs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high VT group (No Intervention)
- Low tidal volume (Experimental)
  Interventions: Procedure: Low tidal volume; Other: low tidal volume

INTERVENTIONS:
Procedure: Low tidal volume — twenty patients were randomly (opaque sealed envelopes) assigned to receive mechanical ventilation in volume-controlled mode either with VT of 10-12 ml/kg predicted body weight (high VT group, n=10) or with VT of 5-7 ml/kg predicted body weight (low VT group, n=10) with an inspiratory fraction of oxygen (FIO2) set at the minimal level at which an arterial oxygen saturation of > 90% and minimal PEEP (4-5cmH2O). The predicted body weight of male patients was calculated as equal to 50+0.91(centimeters of height-152.4); that of female patients was calculated as equal to 45.5+0.91(centimeters of height-152.4).
  Arms: Low tidal volume
Procedure: Low tidal volume — Immediately after ICU admission, once all inclusion and exclusion criteria were met and consent obtained, twenty patients (16 men, 4 women, median age of 49 yrs) were randomly (opaque sealed envelopes) assigned to receive mechanical ventilation in volume-controlled mode either with VT of 10-12 ml/kg predicted body weight (high VT group, n=10) or with VT of 5-7 ml/kg predicted body weight (low VT group, n=10) with an inspiratory fraction of oxygen (FIO2) set at the minimal level at which an arterial oxygen saturation of > 90% and minimal PEEP (4-5cmH2O). The predicted body weight of male patients was calculated as equal to 50+0.91(centimeters of height-152.4); that of female patients was calculated as equal to 45.5+0.91(centimeters of height-152.4)
  Arms: Low tidal volume
Other: low tidal volume — tidal volume of 5-7 ml/kg predicted body weight
  Arms: Low tidal volume

SUMMARY:
Objective: To compare the effects of a protective versus a conventional ventilatory strategy, on systemic and in lung production of tumor necrosis factor-alpha (TNF-alpha) and interleukin-8 (IL-8) in patients without lung disease.

Hypothesis: High tidal volumes induce inflammation in patients without lung disease Design: Prospective control-randomized study. Patients and Setting: Twenty patients without lung disease and submitted to mechanical ventilation admitted to one trauma and one general adult intensive care unit of two different university hospitals.

Interventions: Patients were randomized to receive mechanical ventilation either with tidal volume (VT) of 10-12 ml/kg predicted body weight (high VT group) or with VT of 5-7 ml/kg predicted body weight (low VT group) with an O2 inspiratory fraction (FIO2) enough to keep arterial oxygen saturation > 90% with positive end-expiratory pressure (PEEP) of 5 cmH2O during 12 hours after admission to the study.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 16 years;
2. anticipated survival > 24 hours;
3. need for mechanical ventilation for at least 12 hours and
4. hemodynamic stability (MAP>65 mmHg, HR<100 beats/min, diuresis > 1 ml/kg/h, no catecholamine requirement or fluid challenge).

Exclusion Criteria:

1. history of any lung disease, use of immunosuppressive medication, recent infections, previous thromboembolic disease, recent ventilatory support, and participation in another clinical trial. Absence of lung disease was defined by the following clinical criteria: (a) no evidence of respiratory infection (white blood cell count <10x103/µl, temperature > 380C, purulent sputum), (b) normal chest roentgenogram, (c) PaO2/FIO2 ratio > 300, (d) and a normal clinical respiratory history.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Lung cytokines in mechanically ventilated patients | 30 months

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Complexo Hospitalar Santa Casa, Porto Alegre, Rio Grande do Sul
  - Hospital de Pronto Socorro, Porto Alegre, Rio Grande do Sul